CLINICAL TRIAL: NCT07287280
Title: A Comparison of the Charlson Comorbidity Index (CCI) vs POSSUM Score for Prediction of Perioperative Complications in Patients Undergoing Oncogynecologic Surgery
Brief Title: Comparing CCI and POSSUM for Predicting Oncogynecologic Surgery Complications
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 339/2568(IRB4); Si 428/2025 (Other: Ethical committee, Faculty of Medicine Sirirak Hospital)
Record Dates: First submitted 2025-06-23; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Surgical Procedures; Risk Assessment; Perioperative Care
Keywords: Gynecologic oncology surgery; Perioperative complications; Charlson comorbidity index; POSSUM; Mortality
MeSH Terms: interventions — Morbidity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CCI score — Charlson comorbidity index included age and medical conditions
  Other Names: Charlson comorbidity index
Other: POSSUM score — POSSUM included physical status and laboratory investigation
  Other Names: Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity

SUMMARY:
With the global rates of gynecologic cancers on the rise, optimizing perioperative care is imperative. Accurate risk prediction is essential for enhancing patient care, directing preoperative interventions, and facilitating informed decision-making in oncology. This research compares two widely-used risk assessment tools: the Charlson Comorbidity Index (CCI) and the Physiological and Operative Severity Score for the enUmeration of Mortality and Morbidity (POSSUM), in predicting perioperative outcomes. The CCI predominantly addresses comorbidities, providing simplicity and broad applicability, while POSSUM incorporates both physiological and operative factors for a more comprehensive risk assessment. Despite their application across various surgical specialties, the specific utility of these tools in onco-gynecologic surgery remains insufficiently explored. The study aims to evaluate the effectiveness of CCI and POSSUM in predicting perioperative complications, with a focus on the incidence of these complications, length of hospital stay, and 30-day mortality. The implementation of these risk tools may enhance multidisciplinary risk management, thus improving patient outcomes in gynecologic oncology surgery.

DETAILED DESCRIPTION:
Onco-gynecologic surgeries, including procedures for ovarian, cervical, uterine, and vulvar cancers, are complex and challenging due to both the technical intricacies of the surgeries and the often compromised health of cancer patients. These procedures carry significant perioperative risks, making optimization of perioperative care critical, especially as global cases of gynecological cancers rise, with millions affected annually. Accurate risk prediction is vital to improve patient outcomes, allowing surgeons and anesthesiologists to tailor preoperative interventions and intraoperative management. These strategies help in identifying high-risk patients, implementing enhanced monitoring, specific anesthetic techniques, or staged surgical approaches to mitigate potential complications.

Two prominent risk assessment tools used in surgical practice are the Charlson Comorbidity Index (CCI) and the Physiological and Operative Severity Score for the enUmeration of Mortality and Morbidity (POSSUM). The CCI, is a weighted index that considers the number and severity of comorbid conditions to predict mortality risk. Its simplicity and reliance on readily available clinical information have led to its widespread adoption in clinical and research settings. Studies have validated its predictive value across various surgical populations, including oncology patients, although its specific utility in onco-gynecologic surgeries needs further exploration.

In contrast, the POSSUM score offers a more comprehensive risk assessment by incorporating both physiological and operative factors. It includes preoperative variables like age and cardiac signs and considers operative factors like procedural complexity and blood loss. This dual approach provides a nuanced prediction of perioperative risk, useful across diverse surgical fields. Despite POSSUM's broad application, its effectiveness specifically in onco-gynecologic surgeries requires additional investigation to fully ascertain its predictive accuracy and utility.

Currently, our center conducts preoperative evaluations involving anesthesiologists and gynecologists, yet formal risk assessments using CCI or POSSUM have not been implemented. Incorporating these tools could enhance multidisciplinary risk management, involving anesthetic teams, ward nurses, gynecologic oncologists, and intensivists. By systematically evaluating patient history, these indices can promote effective interdisciplinary communication, significantly improve patient safety, and optimize surgical outcomes.

This study aims to compare CCI and POSSUM in predicting perioperative complications, including both anesthetic and surgical complications in onco-gynecologic surgery. Additionally, it seeks to report the incidence of complications, length of hospital stay, and 30-day mortality, providing valuable insights into optimizing patient care in this challenging field.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient underwent elective onco-gynecologic surgery

Exclusion Criteria:

* Patient required emergency surgery from any indication
* Patient chart that not contained primary outcome data eg. absent of the anesthetic record

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged >,= 18 years, underwent elective onco-gynecologic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of CCI and POSSUM to predict perioperative complications | from the date of starting surgery to the date of hospital discharge, up to 30 days
  To compare the prediction of perioperative anesthetic and surgical morbidity by the Charlson-Comorbidity Index versus POSSUM score in patients undergoing elective onco-gynecological surgery

SECONDARY OUTCOMES:
Intraoperative hypotension | Within 24 hours from starting of surgery
  Intraoperative complications related to anesthesia: intraoperative hypotension
Quantity of intraoperative blood loss | Within 24 hours from starting of surgery
  Intraoperative blood loss estimated by anesthetic personnel
Rate of blood transfusion | Within 24 hours from starting of surgery
  Intraoperative rate and amount of packed red cells blood transfusion and/or blood component
Rate of vasopressor usage | from the time staring of surgery to the time of finishing surgery, up to 12 hours
  Intraoperative rate and amount of vasopressor usage
Clavian-Dindo classification of surgical complications | from the date of starting surgery to the date of hospital discharge, up to 30 days
  Rate of surgical complications using Clavian-Dindo classification of surgical complications Grade 1 Treatment with simple medication Grade 2 Others medications from grade 1 Grade 3a Surgical intervention under local/regional anesthesia Grade 3b Surgical intervention under general anesthesia Grade 4a Need ICU with single organ dysfunction Grade 4b Need ICU with multiple organ dysfunction Grade 5 Death
ICU admission | within 24 hours postoperative
  Rate of intensive care unit admission in the postoperative period
Reoperation | within 24 hours postoperative
  Rate of reoperation
Myocardial infarction or myocardial injury | from the date of starting surgery to the date of hospital discharge, up to 30 days
  Rate of postoperative myocardial infarction and myocardial injury after non-cardiac surgery (MINS)defines as an >1 fold-elevated cTn (>99th percentile of the upper reference limit) of presumed ischemic origin (excluding nonischemic etiologies such as pulmonary embolism, stroke, and sepsis) and is associated with adverse short- and long-term outcomes. (from the 2024 AHA/ACC/ACS/ASNC/HRS/SCA/ SCCT/SCMR/SVM Guideline for Perioperative Cardiovascular Management for Noncardiac Surgery: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines)
Acute kidney injury | from the date of starting surgery to the date of hospital discharge, up to 30 days
  Rate of acute kidney injury which defined follow the KDIGO clinical practice guidelines for acute kidney injury 2020
Postoperative pulmonary complications | from surgery from the date of starting surgery to the date of hospital discharge, up to 30 days
  Rate of postoperative pulmonary complications which defined follow the European Perioperative clinical outcome (EPCO) definition for postoperative pulmonary complications
Mortality rate | From the day of surgery to 30 days post operation
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data supporting the findings of this study are available upon reasonable request, subject to approval and permission from the hospital's director.